CLINICAL TRIAL: NCT00057707
Title: Randomized, Double-Blinded, Placebo Controlled Study of the Effects of Modafinil on Cognitive Function in Patients With Schizophrenia and Normal Controls Based on COMT Genotype
Brief Title: Effects of Modafinil on Brain Function in Patients With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Purpose: Other
Other Study IDs: 030143; 03-M-0143
Record Dates: First submitted 2003-04-05; First posted 2003-04-07 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2017-06-16

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Catecholamines; Dopamine; fMRI; Working Memory; Clinical Trial; Stabilization; Inpatients; Placebo; Modafinil; Normal Volunteers; Schizophrenia; Schizoaffective Disorder; Healthy Volunteer; HV
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Modafinil; Neuropsychological Tests

INTERVENTIONS:
Drug: Modafinil — Placebo 1 week-Wash out 1 week - Drug 1 week (or vice versa)
Procedure: Functional MRI
Procedure: Neuropsychological Testing

SUMMARY:
This study will evaluate whether modafinil improves cognition in patients with schizophrenia and healthy volunteers. Modafinil is a drug that has been FDA approved for day-time sleepiness and allegedly increase the amount of the neurotransmitter dopamine in the frontal cortex of the brain

...

DETAILED DESCRIPTION:
Psychopharmacological modulation of the catecholaminergic system can enhance some aspects of cognitive function. For example, COMT inhibitors can slightly improve working memory/executive function. Similarly, modafinil, a catecholaminergic agonist that increases extracellular dopamine in the prefrontal cortex was also shown to improve delay-dependent working memory. Differences in the response between individuals might be related to a number of factors, including variations in the genes. The recent finding that a polymorphism in the catechol-o-methyl-transferase (COMT) gene, which produces a 4 fold change in enzyme activity, accounts for 4% of the variance in performance of working memory tasks in humans suggest that COMT genotype may predict response to COMT inhibitors or to other agonists that increase catecholaminergic function in the frontal cortex.

In the present investigation our goal is to examine, in normal controls and patients with schizophrenia, the effect of modafinil, a drug that increases DA output in the frontal cortex, on cognitive function and brain physiology. We predict that both normal controls and patients with schizophrenia with the val/val genotype will have a significant improvement in working memory compared with individuals possessing other genotypes. Furthermore, in conjunction with other NIMH imaging protocols, we predict that modafinil will produce a similar genotype-dependent effect on the neurophysiological correlates related to working memory assayed with fMRI. The present protocol will provide new insights on the importance of this genetic polymorphism in the regulation of aminergic-controlled cognitive function in normal individuals. Furthermore, this protocol will test whether modafinil offers a new treatment -based on genotype - for cognitive impairment in schizophrenia. The FDA granted a waiver for the use of Modafinil in this study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Prior participation under NIH protocol # 95-M-0150, or new normal volunteers. Patients with Schizophrenia or Schizoaffective disorder that meet criteria for NIH protocol # 95-M-0150 will be included.

No active Axis I or Axis II diagnosis in normal volunteers.

Age range: 18-50 years.

EXCLUSION CRITERIA:

Subjects with a history of cardiovascular disease, liver disease and other medical illnesses, current active substance abuse or history of substance abuse for more than 5 years, and untreated or uncontrolled hypertension will be excluded. Individuals with persistent tardive dyskinesia will be excluded from the study. An electrocardiogram, blood pressure, pulse rate and metabolic panel including LFTs will be checked on all subjects prior to participation in the study.

Schizophrenic patients taking, a COMT inhibitor, buproprion, stimulants, other cognitive enhancers or any illicit drugs of abuse, or MAO inhibitors will be excluded.

Normal control subjects taking any medications affecting brain function will be excluded.

Pregnant or breastfeeding women. Women of childbearing potential will undergo a urine pregnancy test the day the study initiates and screened by history for the possibility of pregnancy.

Patients with significant history of violence against self or others as established in protocol # 89-M-0160 (Inpatient Evaluation of Neuropsychiatric Patients)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 176 (Actual)
Dates: Start 2003-03-26; Primary Completion 2017-06-16 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
Genetic differences in working memory testing or fMRI activation

SECONDARY OUTCOMES:
Panss, Ham-A, Blood draws for drug levels and liver enzymes

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Apud, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Aguirre JA, Cintra A, Hillion J, Narvaez JA, Jansson A, Antonelli T, Ferraro L, Rambert FA, Fuxe K. A stereological study on the neuroprotective actions of acute modafinil treatment on 1-methyl-4-phenyl-1,2,3,6-tetrahydropyridine-induced nigral lesions of the male black mouse. Neurosci Lett. 1999 Nov 19;275(3):215-8. doi: 10.1016/s0304-3940(99)00706-5. PMID 10580713
- [Background] Aksoy S, Klener J, Weinshilboum RM. Catechol O-methyltransferase pharmacogenetics: photoaffinity labelling and western blot analysis of human liver samples. Pharmacogenetics. 1993 Apr;3(2):116-22. doi: 10.1097/00008571-199304000-00008. PMID 8518836
- [Background] Andreasen NC, Arndt S, Cizadlo T, O'Leary DS, Watkins GL, Ponto LL, Hichwa RD. Sample size and statistical power in [15O]H2O studies of human cognition. J Cereb Blood Flow Metab. 1996 Sep;16(5):804-16. doi: 10.1097/00004647-199609000-00005. PMID 8784225